CLINICAL TRIAL: NCT00859989
Title: Obesity Reduction Black Intervention Trial (ORBIT)
Brief Title: A Weight-Loss Program in Helping Obese Black Women Lose Weight
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Marian Fitzgibbon, University of Illinois Cancer Center
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000635687; UIC-2004-0748
Record Dates: First submitted 2009-03-10; First posted 2009-03-11 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer; Obesity; Weight Changes
Keywords: breast cancer; weight changes; obesity
MeSH Terms: conditions — Breast Neoplasms; Obesity; Body Weight Changes | interventions — Counseling; Early Intervention, Educational; Immunoenzyme Techniques

INTERVENTIONS:
Behavioral: behavioral dietary intervention
Behavioral: exercise intervention
Behavioral: telephone-based intervention
Other: counseling intervention
Other: educational intervention
Other: immunoenzyme technique
Other: laboratory biomarker analysis
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: evaluation of cancer risk factors
Procedure: support group therapy

SUMMARY:
RATIONALE: A diet and physical activity program followed by a weight-loss maintenance program may help obese black women lose weight. It is not yet known whether a weight-loss program is more effective than a general health education program in helping obese black women lose weight. Weight loss may reduce a person's risk of developing cancer.

PURPOSE: This randomized phase III trial is studying a weight-loss program to see how well it works in helping obese black women lose weight.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the effectiveness of a 24-week diet and physical activity intervention and a 1-year maintenance intervention designed to produce and maintain weight loss in obese black women.
* To estimate the effect of these interventions on changes in fasting serum insulin, glucose, and free IGF-1, IGFBP-1, and IGFBP-2 levels as well as total IGF-1 and IGFBP-3 levels.

Secondary

* To compare changes in dietary consumption of total calories, total fat, fruits, vegetables, and fiber as well as physical activity in participants undergoing a weight-loss intervention vs a control intervention.
* To compare changes in knowledge, attitudes, self-efficacy, and social support related to diet, physical activity, and weight loss in participants undergoing a weight-loss intervention vs a control intervention.
* Assess the efficacy of a weight-loss intervention mechanism and the association between weight loss and weight loss maintenance with potential biologic mediators of breast cancer risk.

OUTLINE: Participants are randomized to 1 of 2 intervention arms.

* Arm I (weight-loss intervention): Participants undergo a combined weight-loss intervention (diet and physical activity) over 24 weeks comprising individualized sessions with an interventionist once monthly and group sessions twice weekly. During the group sessions, participants receive information about diet, physical activity, and weight loss and take part in exercise classes. Participants receive handouts, food-measuring tools, and pedometers. Participants also discuss goal setting and problem solving. During the individualized sessions, participants undergo motivational interviewing (MI) to assess their individual needs and to motivate them to make or sustain behavioral changes.

Beginning 1 month after completion of the combined weight-loss intervention, participants undergo a weight-loss maintenance intervention over 12 months. Participants continue their exercise classes twice weekly and receive a copy of the aerobic exercise class videotape for use at home. Prior to each exercise session, participants may share their weight-loss experiences (e.g., successes, struggles) or a motivational or informational story, article, or prayer with other group members. Participants also receive weekly newsletters that include information presented in the original weight-loss intervention, opportunities in the community for physical activity (e.g., ice skating, swimming, or local walks), and further advice on maintaining weight loss. Participants undergo 4 MI sessions over the telephone that address diet, physical activity, and weight-loss maintenance strategies. The MI sessions also provide an opportunity for individualized problem solving.

* Arm II (control intervention): Participants undergo a control intervention over 24 weeks comprising weekly newsletters on general health topics, such as first aid, smoking cessation, cancer screening, and disease prevention, and monthly general health classes that demonstrate information conveyed in the newsletter (e.g., first-aid techniques).

After completion of the control intervention, participants undergo a control maintenance intervention over 12 months comprising a monthly newsletter on general health topics. After completion of the maintenance intervention, participants undergo 10 intervention sessions and receive the same study-related materials (handouts, food-measuring tools, and pedometers) as in arm I.

Blood samples are collected at baseline, 24 weeks, and 18 months for laboratory biomarker studies. Samples are analyzed for insulin levels by radioimmunoassay, glucose concentrations, and total and free IGF-1, IGFBP-1, IGFBP-2, and IGFBP-3 by enzyme-linked immunoassay.

Participants complete questionnaires at baseline, 24 weeks, and 18 months to assess diet, physical activity, cognitive measures (attitudes, beliefs, and self-efficacy), social support, and environmental measures.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Self-identified as Black or African-American
* Body mass index ≥ 30 kg/m²

PATIENT CHARACTERISTICS:

* Pre- or perimenopausal
* Not pregnant or nursing
* Not planning to become pregnant
* Not planning to move from the Chicago area during the active and maintenance study interventions (18 months)
* No exercise intolerance due to chronic obstructive pulmonary disease (e.g., emphysema, chronic bronchitis, or exercise-induced asthma)
* No cancer requiring treatment within the past 5 years, except nonmelanoma skin cancer
* No diabetes
* No uncontrolled hypertension

  * Participants on hypertensive medication may be eligible upon approval by the Investigator
* None of the following conditions:

  * Unstable angina
  * Orthostatic hypotension
  * Moderate to severe aortic stenosis
  * Uncontrolled arrhythmia
  * Uncontrolled congestive heart failure
  * Pulmonary embolism within the past 6 months
  * History of cardiac arrest
* No significant mental illness (e.g., schizophrenia or unmedicated bipolar disorder)
* No alcohol intake of > 2 drinks per day
* No illegal drug use
* No laxative abuse (i.e., > twice the recommended dose)

PRIOR CONCURRENT THERAPY:

* No concurrent treatment for an eating disorder
* No concurrent medications (e.g., hormone-replacement therapy) that could interfere with adherence to an exercise program or could interfere with study outcomes
* No concurrent participation in a formal weight-loss program
* No concurrent pharmacotherapy for weight loss

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2004-07; Primary Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Body mass index as assessed at baseline, 24 weeks, and 18 months
Changes in glucose, insulin, and IGF levels as assessed at baseline, 24 weeks, and 18 months

SECONDARY OUTCOMES:
Changes in diet and physical activity as assessed by Block 98 FFQ and Stanford 7-Day Physical Activity Recall questionnaires at baseline, 24 weeks, and 18 months
Changes in knowledge, attitudes, self-efficacy, and social support related to diet, physical activity, and weight loss as assessed by Nutrition Attitudes Scale, Self-Efficacy for Eating and Exercise Behaviors, and Social Support for Eating and Exerci ...

CONTACTS AND LOCATIONS:
Overall Officials: Marian Fitzgibbon, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Cancer Center, Chicago, Illinois, United States